CLINICAL TRIAL: NCT02501759
Title: Pilot Study of Transrectal Multiparametric MRI-Guided Biopsy: Role in Prostate Cancer Evaluation
Brief Title: Transrectal MRI-Guided Biopsy in Identifying Cancer in Patients With Suspected Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment and funding loss.
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Medical Research Foundation, Oregon (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Fergus Coakley, Professor and Chair, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00010086; NCI-2015-00930 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SOL-13142-LM; IRB00010086 (Other: OHSU Knight Cancer Institute); P30CA069533 (NIH)
Record Dates: First submitted 2015-07-15; First posted 2015-07-17 (Estimated); Results first posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Health Status Unknown; Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gadodiamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (MRI, MRI-guided biopsy, TRUS-guided biopsy) (Experimental): Patients receive gadodiamide IV and undergo a diagnostic multiparametric endorectal MRI. Patients with lesions visible on the diagnostic multiparametric endorectal MRI undergo transrectal MRI-guided biopsy within 2 weeks of diagnostic multiparametric endorectal MRI. Patients then undergo TRUS-guided biopsy per standard clinical care approximately 2 weeks after transrectal MRI-guided biopsy.
  Interventions: Procedure: 3 Tesla Magnetic Resonance Imaging; Radiation: Gadodiamide; Procedure: Multiparametric Magnetic Resonance Imaging; Procedure: Transrectal Biopsy; Procedure: Ultrasound-Guided Prostate Biopsy

INTERVENTIONS:
Procedure: 3 Tesla Magnetic Resonance Imaging — Undergo diagnostic multiparametric endorectal MRI with gadodiamide contrast
  Other Names: 3 Tesla MRI; 3T MRI
Radiation: Gadodiamide — Given IV
  Other Names: DV 7572; Gadolinium-DTPA-BMA; Gd-DTPA-BMA; HSDB 7547; OmniScan
Procedure: Multiparametric Magnetic Resonance Imaging — Undergo diagnostic multiparametric endorectal MRI with gadodiamide contrast
  Other Names: Multiparametric MRI
Procedure: Transrectal Biopsy — Undergo transrectal MRI-guided biopsy
  Other Names: Transrectal Prostate Biopsy
Procedure: Ultrasound-Guided Prostate Biopsy — Undergo TRUS-guided biopsy

SUMMARY:
This pilot clinical trial studies transrectal magnetic resonance imaging (MRI)-guided biopsy to see how well it works in identifying cancer in patients with suspected prostate cancer who are scheduled to undergo standard biopsy. Transrectal MRI-guided biopsy uses a thin needle inserted through the rectum into the prostate and takes a sample of tissue, guided by MRI. MRI uses magnets to take pictures of the prostate and may be able to identify cancer. Transrectal MRI-guided biopsy may be more accurate and cause patients less pain than standard ultrasound-guided biopsy. It is not yet known whether transrectal MRI-guided biopsy is more effective than ultrasound-guided biopsy in identifying prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To improve the treatment of patients with prostate cancer utilizing diagnostic multi-parametric magnetic resonance imaging (MRI) and MRI-guided prostate biopsy combined with molecular and clinical data to help determine the extent of prostate cancer and risk of disease progression.

II. To determine the relative accuracy of transrectal MRI-guided versus ultrasound-guided biopsy for the diagnosis of prostate cancer in patients with an appropriate dominant target lesion at multiparametric MRI, using pooled cancer diagnoses by either MRI-guided or ultrasound-guided biopsy as the reference standard.

III. To determine the proportion of positive transrectal MRI-guided biopsies that demonstrate a higher Gleason score than contemporaneous transrectal ultrasound guided biopsy.

IV. To determine the management impact of transrectal MRI-targeted biopsy results as compared to transrectal ultrasound (TRUS)-guided systematic biopsy results.

OUTLINE:

Patients receive gadodiamide intravenously (IV) and undergo a diagnostic multiparametric endorectal MRI. Patients with lesions visible on the diagnostic multiparametric endorectal MRI undergo transrectal MRI-guided biopsy within 2 weeks of diagnostic multiparametric endorectal MRI. Patients then undergo TRUS-guided biopsy per standard clinical care approximately 2 weeks after transrectal MRI-guided biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled TRUS-guided biopsy because of clinically suspected prostate cancer (abnormal serum prostate-specific antigen [PSA] level and/or abnormal digital rectal examination)
* No treatment for prostate cancer has been administered or will be administered before TRUS guided biopsy
* Patient willing to undergo scheduled standard of care TRUS guided biopsy
* Patient willing and able to provide written informed consent, including willingness to undergo both endorectal multiparametric MRI and transrectal MRI-guided biopsy at Oregon Health & Science University (OHSU)
* Laboratory values and anticoagulation management per consensus guidelines, including:
* International normalized ratio (INR) >= 1.5
* Platelets >= 50,000

Exclusion Criteria:

* Known contraindication to MRI (e.g., severe claustrophobia, intracranial aneurysm clips, intraocular metallic foreign body, cardiac pacemaker); an extensive screening questionnaire will be completed by the subject as part of standard OHSU MRI safety measures
* Known contraindication to intravenous gadolinium contrast administration (e.g., renal impairment, known allergy); standard institutional policies on gadolinium and renal function will be followed
* Contraindication to placement of endorectal MRI coil, biopsy device or ultrasound probe (e.g., severe hemorrhoids, anal fissure, recent rectal surgery, or prior abdominoperineal resection)
* Previous inclusion in the study (e.g., a patient who has had negative TRUS and MRI-guided biopsies but continues to have a rising PSA)
* Active urinary tract infection
* Member of vulnerable population including prisoners or mentally disabled patients, in accordance with U.S. Department of Health and Human Services (DHHS) definitions

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12-31 (Actual); Study Completion 2017-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fergus Coakley, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (MRI, MRI-guided Biopsy, TRUS-guided Biopsy)
Started | 2
Completed | 1
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (MRI, MRI-guided Biopsy, TRUS-guided Biopsy)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of MRI-guided Biopsies That Demonstrate a Higher Gleason Score Than Contemporaneous TRUS Guided Biopsy
Description: The proportion of MRI-guided biopsies that demonstrate a higher Gleason score than contemporaneous TRUS guided biopsy for all patients diagnosed of prostate cancer based on the reference standard will be estimated. McNemar's test will be used to assess whether the MRI-guided biopsies are more likely to yield a higher Gleason score compared with TRUS guided biopsy. Simple logistic regression model will be used to assess the association between the higher Gleason score and patient characteristics and/or clinical information for patients diagnosed of prostate cancer.
Time Frame: Up to 42 days (6 weeks)
Population: Due to low enrollment, insufficient data was collected to report this outcome
Arm/Group | Diagnostic (MRI, MRI-guided Biopsy, TRUS-guided Biopsy)
Number analyzed (Participants) | 0

2. Primary Outcome: Sensitivity of MRI-guided Biopsy
Description: The presence of cancer on either biopsy or absence of cancer on both will be used as the reference standard. For comparison of the two methods, the 2X2 matched sample tables will be presented, and the difference in sensitivity estimated. The relative accuracy of MRI- versus TRUS-guided biopsy will be compared using McNemar's test. To explore potential associations between the accuracy of each method with patient characteristics and/or clinical information, a binary endpoint will be created to reflect agreement between each method and the reference standard.
Time Frame: Up to 2 weeks after diagnostic MRI
Population: Due to low enrollment, insufficient data was collected to report this outcome
Arm/Group | Diagnostic (MRI, MRI-guided Biopsy, TRUS-guided Biopsy)
Number analyzed (Participants) | 0

3. Primary Outcome: Sensitivity of TRUS-guided Biopsy
Description: as for outcome 2
Time Frame: Up to 2 weeks after MRI-guided biopsy
Population: Due to low enrollment, insufficient data was collected to report this outcome
Arm/Group | Diagnostic (MRI, MRI-guided Biopsy, TRUS-guided Biopsy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Diagnostic (MRI, MRI-guided Biopsy, TRUS-guided Biopsy)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Since recruitment was very low and funding did not materialize, the study was closed early and insufficient data was collected to analyze and report the outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes